CLINICAL TRIAL: NCT05266209
Title: Comparison of Coconut and Sunflower Oil Application in Preserving Skin Integrity of Infants in Neonatal Intensive Care Unit
Brief Title: Comparison of Coconut and Sunflower Oil Application in Preserving Babies' Skin Integrity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, öznur tiryaki, Nurse, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0
Record Dates: First submitted 2022-02-02; First posted 2022-03-04 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Skin Care
Keywords: Coconut oil; Sunflower oil; neonatal; Neonatal Intensive Care Unit; skin care

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Masking Description: The researcher is not blind since the group of infants will be assigned by the researcher in order. The statistician was also blinded for the data analysis purpose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental (coconut oil group) (Experimental): Before moistening, the skin of newborns is evaluated using the Newborn Skin Condition Evaluation Form form.
  Moisturizers are applied to the thorax, back, arms and legs by massage, respectively, and the skin is absorbed. If it is to be applied for the first time, it is applied to a small area of the body under the control of a doctor. If there is no reaction, it is applied by massaging other areas. Since the babies to be included in the sample group are borderline and moderately premature (34-37W), 3-4 ml/kg (coconut oil)moisturizer will be applied.
  Evaluation with NSCE form: Evaluations will be made using the NSCE form 48-72 hours after each application (Monday, Thursday, Sunday). Routine care will be applied to the skin of the newborns in the control group in the hospital. The control group will be evaluated using the NSCE form 3 days a week (Monday, Thursday, Sunday).
  Interventions: Other: Coconut oil skin care group
- Experimental (sunflower oil group) (Other): Before moistening, the skin of newborns is evaluated using the Newborn Skin Condition Evaluation Form form.
  Moisturizers are applied to the thorax, back, arms and legs by massage, respectively, and the skin is absorbed. If it is to be applied for the first time, it is applied to a small area of the body under the control of a doctor. If there is no reaction, it is applied by massaging other areas. Since the babies to be included in the sample group are borderline and moderately premature (34-37W), 3-4 ml/kg (sunflower oil) moisturizer will be applied.
  Evaluation with NSCE form: Evaluations will be made using the NSCE form 48-72 hours after each application (Monday, Thursday, Sunday).
  Interventions: Other: Coconut oil skin care group
- No Intervention (Control group) (No Intervention): Before moistening, the skin of newborns is evaluated using the Newborn Skin Condition Evaluation Form form.
  Routine maintenance of the intensive care unit will be implemented. Evaluation with NSCE form: Evaluations will be made using the NSCE form 48-72 hours after each application (Monday, Thursday, Sunday). Routine care will be applied to the skin of the newborns in the control group in the hospital. The control group will be evaluated using the NSCE form 3 days a week (Monday, Thursday, Sunday)

INTERVENTIONS:
Other: Coconut oil skin care group — No special technique was used for sample selection, random sample selection will be made. In the evaluation made according to the large effect size, the number of samples determined for Power: 0.80, :0.20 and :0.05 was determined as 66, with a minimum of 22 for each group. Calculations were made in computer environment using Power analysis (G*Power 3.1.9.2) program. Random selection method will be used while creating research groups. Coconut oil, sunflower oil and control groups will be formed according to the order of admission to the unit. E.g; Coconut oil is planned for the first hospitalized newborn, sunflower oil for the second newborn, and third hospitalized newborn control group. This order will be repeated until a sufficient number of cases is reached when the newborns are included in the groups.
  Other Names: sunflower oil skin care group
  Arms: Experimental (coconut oil group); Experimental (sunflower oil group)

SUMMARY:
This study was planned to examine the effects of coconut and sunflower oils applied to the skin of newborns on the daily fluid intake and output of the baby, the weight gain/decrease status and skin integrity.

DETAILED DESCRIPTION:
Although there is no consensus on the use of products in daily skin care to maintain the skin integrity of newborns, many products are used. These products; mustard, sunflower, sesame, coconut, olive, soybean, palm oils, ointment (Auqophor), cream (Eucerin) and moisturizers. It is stated that these products prevent skin drying and fissures, maintain skin integrity, and reduce transepidermal fluid loss (Vaseline).

Sunflower oil accelerates the maturation of the skin barrier, there is less weight loss in newborns younger than 35 weeks of gestation who are massaged with sunflower oil compared to the control group, the incidence of nosocomial infections in newborns who receive skin care with sunflower oil is lower than the control group, sunflower oil protects the newborn from infections, olive oil, more effective than oils such as soybean oil and mustard oil; In another study, it was determined that skin care applied to preterm newborns with sunflower oil reduced mortality by 26%, the duration of hospitalization was shorter in newborns treated with sunflower oil than the control group, and regular use of moisturizers had no effect on the incidence of infection. Recently, it has been reported that topical application of coconut oil is safe and feasible in very preterm infants and has beneficial effects on skin condition and recovery of infants. In a systematic review of randomized studies evaluating the effects of topical coconut oil in preterm infants, it was emphasized that in general, transepidermal fluid loss and infection rate were reduced in infants in the coconut oil group, the growth and skin integrity of the infants were better, and no significant side effects were experienced. In a study comparing coconut and carrot oils, it was stated that the skin flora and barrier function were better in babies using coconut oil.

Comparison of the application of Coconut and Sunflower Oil in the preservation of skin integrity, the amount of fluid ingested/extracted daily, and weight gain/decrease in infants hospitalized in the Neonatal Intensive Care Unit.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary verbal and written consent of the parents of the newborn,
* The gestational week of the newborn is 34 and above,
* The birth weight of the newborn is 2000 g and above,
* The hospitalization of the newborn is the first day of birth.

Exclusion Criteria:

* Unstable clinical condition and vital signs,
* Having a major congenital anomaly,
* High risk of infection due to surgery,
* More than 5% of the body surface is a skin disease,
* External application of medication to the skin in its treatment.

Ages: 34 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
effect on skin integrity | Evaluation with Newborn Skin Condition Evaluation Form (NSCE) form: Evaluations will be made using the YCDD form 48-72 hours after each application (Monday, Thursday, Sunday).
  Evaluation with Newborn Skin Condition Evaluation Form (NSCE) form: Evaluations will be made using the YCDD form 48-72 hours after each application (Monday, Thursday, Sunday).
  Skin condition scoring of the newborn; It is performed according to the presence of signs of redness, dryness and deterioration of skin integrity/peeling. It was developed in a three-point Likert format and each item/finding is given a score from 1 to 3. The lowest score that can be obtained as a result of the evaluation is 3, and the highest score is 9. A total score higher than 3 indicates that there is a risk of deterioration of the skin integrity of the newborn, while a high score indicates that the newborn's skin condition is poor.
the effect of the baby's weight gain/decrease on 7,14, 21, 28 days | The scale is sensitive enough to measure in very small units.
  The baby's weight will be measured on days 7, 14, 21, 28, naked and without diapers.

CONTACTS AND LOCATIONS:
Overall Officials: NURSAN ÇINAR, Prof, Principal Investigator — Sakarya University; HAMİDE ZENGİN, Asis Prof, Principal Investigator — Bilecik Seyh Edebali Universitesi; İBRAHİM CANER, Prof, Principal Investigator — Sakarya University; ERTUĞRUL GÜÇLÜ, Prof, Principal Investigator — Sakarya University; ÖZNUR TİRYAKİ, PhD, Principal Investigator — Sakarya Education and Research Hospital; MELTEM KARABAY, Asis Prof, Study Chair — Sakarya University
Locations (1):
- Sakarya Education and Training Hospital, Sakarya, Adapazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No